CLINICAL TRIAL: NCT04202393
Title: RCT to Improve Post-Hospital Treatment Adherence for Comorbid Substance Use and Bipolar Disorders
Brief Title: Intervention for Comorbid Substance Use and Bipolar Disorders
Acronym: ITAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1370188-2; R01MH122870 (NIH)
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Disorder; Substance Use Disorders
MeSH Terms: conditions — Bipolar Disorder; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Treatment Adherence Program (ITAP) (Experimental): A combination of in-person and phone sessions along with significant other involvement over 6 months post-hospitalization.
  Interventions: Behavioral: Integrated Treatment Adherence Program (ITAP)
- Safety Assessment and Follow-up Evaluation (SAFE) (Active Comparator): Enhanced symptom monitoring and safety evaluation over 6 months post-hospitalization.
  Interventions: Behavioral: Safety Assessment and Follow-up Evaluation (SAFE)

INTERVENTIONS:
Behavioral: Integrated Treatment Adherence Program (ITAP) — Psychosocial support and treatment to improve treatment adherence, symptoms, and functioning.
  Arms: Integrated Treatment Adherence Program (ITAP)
Behavioral: Safety Assessment and Follow-up Evaluation (SAFE) — Enhanced assessment and evaluation with clinician feedback.
  Arms: Safety Assessment and Follow-up Evaluation (SAFE)

SUMMARY:
This trial aims to evaluate the effectiveness of a novel intervention for patients with co-occurring bipolar and substance use disorders following a psychiatric hospitalization. Half of the participants will receive a specialized psychosocial intervention program, while the other half will receive an enhanced safety monitoring program, both provided in addition to their routine care.

ELIGIBILITY:
Inclusion:

* Diagnosis of a bipolar-spectrum disorder
* Diagnosis of a substance use disorder
* Taking at least one mood-stabilizing medication

Exclusion:

* Unable to speak and read English
* Younger than age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Clinician Rating (QIDS-C) | 6 months
  The Quick Inventory of Depressive Symptomatology - Clinician Rating (QIDS-C) assesses depressive symptom severity. Total scores range from 0 to 27 and higher scores indicated higher symptom severity.
Clinician-Administered Rating Scale for Mania (CARS-M) | 6 months
  The Clinician-Administered Rating Scale for Mania (CARS-M) assesses mania symptom severity. Total scores range from 0 to 50 and higher scores indicated higher symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital; Ivan Miller, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Upload to NIMH Data Archive